CLINICAL TRIAL: NCT03623724
Title: i-Care for Depression: Blending Face-to-face Psychotherapy With Internet and Mobile Digital Solutions
Brief Title: iCare4Depression: Effectiveness of a Blended Cognitive-Behavioral Therapy in Routine Practice
Acronym: iCare4Dep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Institute of Maia (Other)
Collaborators: INESC TEC (Unknown); University of Limerick (Other); VU University of Amsterdam (Other); Center of Psychology at University of Porto (Unknown); ARS - Norte (Unknown)
Responsible Party: Principal Investigator, João Salgado, Assistant Professor, University Institute of Maia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTDC/MHC-PCL/1991/2014
Record Dates: First submitted 2018-07-24; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Major Depression
Keywords: Major Depression; Blended Therapy; Randomized Clinical Trials; e-Mental Health; Routine Practice
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The RCT is composed by an experimental condition and a control condition. In the experimental condition, patients will receive a treatment that integrates face-to-face cognitive-behavioral sessions with online sessions delivered through Moodbuster system (bCBT). In the control condition, patients will receive TAU that consists in routine care that they usually receive in primary care. We will not interfere with treatments delivered in TAU, but the intervention will be tracked, as well as medicine intake. One-hundred patients will be recruited and randomized in two conditions: 50 for bCBT condition and 50 for TAU condition. New cases of Major Depression signaled by GPs or other healthprofessionals will be invited to participate in the RCT. Once obtained the signed informed consent, the patients will be randomized at an individual level. The allocation will be performed by an independent researcher not involved in data collection using an automated computer-based random intergenerator.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blended Cognitive-behavioral Therapy (Experimental): The experimental condition refers to a blended treatment that integrates empirically-supported face-to-face cognitive-behavioral psychotherapy with a mobile phone application and a web platform - blended cognitive-behavioral therapy (bCBT). The intervention includes ten face-to-face cognitive-behavioral sessions combined with nine online sessions based on the self-help treatment modules of the Moodbuster (psychoeducation, exercise therapy, behavioral activation, problem solving, cognitive restructuring and relapse prevention) delivered over a period of 16 weeks. 50 patients will be integrated in this experimental condition.
  Interventions: Behavioral: blended Cognitive-behavioral Therapy
- Treatment-As-Usual (Active Comparator): The control condition concerns the treatment-as-usual (TAU) that consists in routine care that patients receive when they are diagnosed with major depression in primary care. We will not interfere with treatments delivered in TAU, but the intervention will be tracked (e.g., medication). The psychiatrist of our team will monitor possible medicine intake (stabilized throughout the trial). 50 patients will be integrated in this condition.
  Interventions: Other: Treatment-As-Usual

INTERVENTIONS:
Behavioral: blended Cognitive-behavioral Therapy — The protocol includes ten face-to-face cognitive-behavioral sessions combined with nine online sessions based on Moodbuster self-help treatment, delivered over a period of 16 weeks. The Moodbuster includes 7 modules (introduction, psychoeducation, behavioral activation, cognitive restructuring, problem solving, exercise and relapse prevention), a calendar and the possibility of sending and receiving messages to and from therapist, respectively. The mobile phone application will be used to support the therapeutic sessions and register the ecological momentary assessments concerning mood, sleep quality, anxiety and other emotional states that will be collected in a daily basis before, during and after the treatment.
  Arms: blended Cognitive-behavioral Therapy
Other: Treatment-As-Usual — The protocol consists in routine care that patients receive when they are diagnosed with major depression in primary care. We will not interfere with treatments delivered in TAU, but the intervention will be tracked (e.g., medication). The psychiatrist of our team will monitor possible medicine intake (stabilized throughout the trial).
  Arms: Treatment-As-Usual

SUMMARY:
The main objective of this research project is to implement and evaluate the clinical effectiveness and cost-effectiveness of a Blended Cognitive-Behavioral Therapy (bCBT) in routine practice, comparing it with Treatment as Usual (TAU). This research project includes a pilot study and a randomized clinical trial (RCT).

The pilot study main objective is to adapt the bCBT based on Moodbuster, an internet-based treatment platform developed by the ICT4Depression Consortium (INESC-TEC, Vrije Universiteit and University of Limerick), to the Portuguese population. More specifically, this pilot study intends: (1) to detect problems and refine procedures, establishing a definitive Portuguese version of the blended treatment; (2) to assess clinical effectiveness (non-controlled), estimating effect sizes at the end of the treatment and follow-up; (3) to assess patients' satisfaction and personal views concerning their process of change; (4) to develop dynamic models of the individual trajectories during treatment based on Ecological Momentary Assessments. The pilot study will involve the participation of psychologists trained in bCBT and 20 participants diagnosed with Major Depression and willing to use the Moodbuster system.

The RCT is composed by two arms (an experimental condition and a control condition) and it will be implemented in routine practice. In the experimental condition, the patients diagnosed with Major Depression will receive a treatment that integrates face-to-face cognitive-behavioral sessions with online sessions available through Moodbuster system (bCBT). In the control condition, patients diagnosed with Major Depression will receive TAU that consists in routine care that patients receive in primary care. The RCT will involve the participation of family doctors and psychologists working in routine practice. One-hundred patients will be recruited and randomized in the two conditions: 50 patients for bCBT condition and 50 patients for TAU condition. The main objectives are: (1) to assess the clinical effectiveness of bCBT and compare it with TAU in routine practice; (2) to estimate and compare cost-effectiveness of both treatments; (3) to assess patients' and clinicians' satisfaction with the bCBT and TAU; (4) to refine the previous models of individual trajectories and to assess differential effects on different patient clusters; (5) to establish guidelines for using bCBT within Portuguese routine practice services.

DETAILED DESCRIPTION:
Internet-based interventions in depression have emerged over the last decades to improve the access to effective treatments. Despite the increasing relevance of these treatments, empirical evidence is still needed to demonstrate their clinical and cost-effectiveness in different healthcare contexts. The present study represents an extension to the Portuguese context of the original trial developed by the ECOMPARED consortium. The overall project involves a pilot study and a randomized clinical trial (RCT).

The pilot study main objective is to adapt the bCBT based on Moodbuster, an internet-based treatment platform developed by the ICT4Depression Consortium (INESC-TEC, Vrije Universiteit and University of Limerick), to the Portuguese population. More specifically, this pilot study intends: (1) to detect problems and refine procedures, establishing a definitive Portuguese version of the blended treatment; (2) to assess clinical effectiveness (non-controlled), estimating effect sizes at the end of the treatment and follow-up; (3) to assess patients' satisfaction and personal views concerning their process of change; (4) to develop dynamic models of the individual trajectories during treatment based on Ecological Momentary Assessments (EMA). The pilot study will involve the participation of psychologists trained in bCBT and 20 participants diagnosed with Major Depression and willing to use the Moodbuster system. The assessment protocol will be implemented at the baseline, during therapeutic sessions, 16 weeks and 26 weeks after baseline and it is composed by several measures that evaluate depressive symptoms, anxiety symptoms, distress, quality of life, working alliance, treatment credibility and expectancy, treatment satisfaction and system usability. Moreover, the EMA concerning mood, sleep quality, anxiety and other emotional states will be collected in a daily basis before, during and after the treatment. The intervention protocol includes ten face-to-face cognitive-behavioral sessions combined with nine online sessions based on the self-help treatment modules of the Moodbuster (psychoeducation, exercise therapy, behavioral activation, problem solving, cognitive restructuring and relapse prevention) delivered over a period of 16 weeks.

The RCT is composed by two arms (an experimental condition and a control condition) and it will be implemented in routine practice. In the experimental condition, the patients diagnosed with Major Depression will receive a treatment that integrates face-to-face cognitive-behavioral sessions with online sessions available through Moodbuster system (bCBT). In the control condition, patients diagnosed with Major Depression will receive TAU that consists in routine care that patients receive in primary care. The RCT will involve the participation of family doctors and psychologists working in routine practice. One-hundred patients will be recruited and randomized in the two conditions: 50 patients for bCBT condition and 50 patients for TAU condition. The main objectives are: (1) to assess the clinical effectiveness of bCBT and compare it with TAU in routine practice; (2) to estimate and compare cost-effectiveness of both treatments; (3) to assess patients' and clinicians' satisfaction with the bCBT and TAU; (4) to refine the previous models of individual trajectories and to assess differential effects on different patient clusters; (5) to establish guidelines for using bCBT within Portuguese routine practice services. The assessment protocol will be implemented at the baseline, during therapeutic sessions, 16 weeks, 26 and 52 weeks after baseline and it is composed by several measures that evaluate depressive symptoms, anxiety symptoms, distress, quality of life, working alliance, treatment credibility and expectancy, treatment satisfaction, system usability and cost-effectiveness. Moreover, the EMA concerning mood, sleep quality, anxiety and other emotional states will be collected in a daily basis before, during and after the treatment. The intervention protocol includes ten face-to-face cognitive-behavioral sessions combined with nine online sessions based on the self-help treatment modules of the Moodbuster (psychoeducation, exercise therapy, behavioral activation, problem solving, cognitive restructuring and relapse prevention) delivered over a period of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years;
* Diagnosis of Major Depression Disorder;
* PHQ-9 score ≥ 9;
* Availability to use the Moodbuster system (online platform and mobile application).

Exclusion Criteria:

* Lack of symptoms for Major Depressive Disorder;
* Lack of proficiency in Portuguese language;
* Not having a computer and/or a smartphone with internet access;
* Presence of severe psychiatric comorbidity requiring alternative treatment, primary to depression treatment;
* High risk of suicide;
* Currently receiving psychotherapy;
* Changes on medication in the last month or plans to change it before the end of the RCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-02 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms from baseline to 52 weeks after baseline | Baseline assessment; therapeutic sessions; 16 weeks after baseline; 26 weeks after baseline; 52 weeks after baseline
  Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001). The PHQ-9 is composed by nine items that assess the severity of the depressive symptoms in a Likert scale of four points (0 = Not at all; 3 = Nearly every day). The total score of this questionnaire can range from 0 to 27 points. A total score between 0 and 4 indicates subclinical symptoms of depression; a total score between 5 and 9 indicates mild depression; a total score between 10 and 14 indicates moderate depression; a total score between 15 and 19 indicates moderately severe depression; and a total score between 20 and 27 indicates severe depression.

SECONDARY OUTCOMES:
Change in the diagnosis of major depression disorder from baseline to 52 weeks after baseline | Baseline assessment; 16 weeks after baseline; 26 weeks after baseline; 52 weeks after baseline
  Structured Clinical Interview for DSM-5 (First, Williams, Karg, & Spitzer, 2015). The diagnostic of Major Depression will be performed by a trained psychologist through the Structured Clinical Interview for DSM-5 (First, Williams, Karg, & Spitzer, 2015). The SCID-5 CV is a structured interview that allows a systematic evaluation of the participants taking into account the classification and diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5; APA, 2013).
Change in the general clinical outcome from baseline to 52 weeks after baseline | Baseline assessment; therapeutic sessions; 16 weeks after baseline; 26 weeks after baseline; 52 weeks after baseline
  Clinical Outcome Routine Evaluation - Outcome Measure (CORE-OM; Evans, Mellor-Clark, Barkham, & Mothersole, 2006). The CORE-OM is a self-report questionnaire composed by 34 items that assess global distress and specific dimensions, namely subjective well-being, problems/symptoms, life functioning and risk/harm. Each item is assessed through a Likert scale of five points (0 = not at all; 4 = most or all the time). The total score of this questionnaire can range from 0 to 136 (this score is obtained by adding the response values of each item). The total mean score is calculated by dividing the total score by the number of completed responses. The mean scores for each dimension are calculated by dividing the total scores by the number of completed item responses for each dimension. Higher scores indicate worse results in terms of global distress, but also for the specific dimensions of the questionnaire.
Change in anxiety symptoms from baseline to 52 weeks after baseline | Baseline assessment; therapeutic sessions; 16 weeks after baseline; 26 weeks after baseline; 52 weeks after baseline
  Generalized Anxiety Disorders (GAD-7; Spitzer, Kroenke, Williams, & Lowe, 2006). The GAD-7 is composed by seven items that assess the symptoms of generalized anxiety in a Likert scale of four points (0 = Not at all; 3 = Nearly every day). The total score ranges from 0 to 21. A total score between 0 and 4 indicates subclinical symptoms of anxiety; a total score between 5 and 9 indicates mild anxiety; a total score between 10 and 14 indicates moderate anxiety; and a total score between 15 and 21 indicates severe anxiety.
Evolution of the working alliance between therapist and patient during therapeutic sessions and follow-up assessments | Therapeutic sessions; 16 weeks after baseline; 26 weeks after baseline; 52 weeks after baseline
  Working Alliance Inventory-Short Revised (WAI-SR; Tracey & Kokotovic, 1989). This questionnaire is composed by 12 items, each one scored in a Likert scale of 5 points (1 = rarely or never; 5 = always). This questionnaire measures three dimensions of the therapeutic alliance, namely: (a) agreement between patient and therapist on the goals of the treatment; (b) agreement between patient and therapist about the tasks to achieve these goals; and (c) the quality of the bond between the patient and therapist. In each dimension the total score can range between 5 and 20, and higher scores indicate better therapeutic alliance.
Usability of the Moodbuster system (web platform and smartphone application) for patients and therapists | 16 weeks after baseline; 26 weeks after baseline; 52 weeks after baseline
  System Usability Scale (SUS; Brook, 1996). The SUS is a self-report scale composed 10 items rated in a Likert scale of five points (1 = completely disagree; 5 = completely agree) to assess the effectiveness, efficiency and satisfaction regarding the Moosbuster system. The total score of this scale can range from 10 to 50 points.
Patients' treatment credibility and expectancy | Baseline assessment
  Credibility and Expectancy Questionnaire (CEQ; Borkovec & Nau, 1972; Devilly & Borkovec, 2000). This questionnaire is composed by two sets of items (some ranging from 1 to 9 and others ranging from 0 to 100%) that assess two separate factors, namely treatment expectancy and rationale credibility. Higher results indicate better patients' credibility and expectancy regarding the treatment.
Patients' treatment satisfaction | 16 weeks after baseline; 26 weeks after baseline; 52 weeks after baseline
  Client Satisfaction Scale (CSQ-8; Larsen, Attkisson, Hargreaves, & Nguyen, 1979). This scale evaluate patients' level of satisfaction with treatment. It is composed of eight items, each one evaluated in a Likert scale of four points (1 = low satisfaction; 4 = high satisfaction). The CSQ-8 is scored by summing the individual item scores. The total score can range from 8 to 32, and high scores indicate greater satisfaction with treatment.
Change in patients' quality of life from baseline to 52 weeks after baseline | Baseline assessment; 16 weeks after baseline; 26 weeks after baseline; and 52 weeks after baseline
  EQ-5D-5L (Brooks & Euroqol Group, 1996). The EQ-5D-5L is a self-report measure that assesses health-related quality of life taking into account five dimensions: (1) mobility, (2) personal care, (3) usual activities, (4) pain/discomfort, and (5) anxiety/depression. Each dimension is rated in 5 levels: (1) no problems, (2) slight problems, (3) moderate problems, (4) severe problems, and (5) extreme problems. A total of 3125 possible health states can be defined by this scale. This health state may be converted into a single index value. Also, it is possible to obtain, through this measure, a quantitative measure of health. The patient can rate their health in a scale ranging between "the best health you can imagine" and "the worst health you can imagine".
Assessment of treatment's cost-effectiveness | Baseline assessment; 16 weeks after baseline; 26 weeks after baseline; and 52 weeks after baseline
  An equivalent measure to Trimbos/iMTA Questionnaires on Costs Associated with Psychiatric Illness (TiC-P; Roijen, van Straten, Donker, & Tiemens, 2002) will be used. This measure, under development, will be used to estimate medical costs and indirect non-medical costs associated with productivity losses due to absenteeism and lower efficiency at work in the last 4 weeks.
Ecological Momentary Assessments | 1 week before treatment, during treatment and 1 week after treatment
  Assessments concerning mood, sleep quality, anxiety and other emotional states that will be collected in a daily basis, in a Likert scale of 7 points.

CONTACTS AND LOCATIONS:
Overall Officials: João Salgado, PhD, Principal Investigator — University Institute of Maia
Locations (1):
- University Institute of Maia, Maia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
The data will be available to other researchers through scientific publications, manuals, books, conferences and other scientific events.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Sousa, M., Barbosa, E., Basto, I., Silva, S., Meira, L., Ferreira, T., & Salgado, J. (2018, April). Blended cognitive-behavioral therapy for depression: The iCare4Depression study protocol. Paper presented at 5th ESRII 2018, Dublin, Ireland. https://docs.wixstatic.com/ugd/1d9a38_aacb4271986d492e8fa1317a6207f077.pdf